CLINICAL TRIAL: NCT05647538
Title: The Effect of Bilateral Uterine Artery Ligation After Intrapartum or Postpartum Hemorrhage on Ovarian Reserve Markers and Pregnancy Outcome
Brief Title: Bilateral Uterine Artery Ligation After Intrapartum or Postpartum Hemorrhage on Ovarian Reserve Markers and Pregnancy Outcome
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ossman, Assistant Professor of Obstetrics and Gynecology Department Tanta, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36034/11/22
Record Dates: First submitted 2022-12-04; First posted 2022-12-12 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Bilateral Uterine Artery Ligation; Intrapartum or Postpartum Hemorrhage; Ovarian Reserve Markers; Pregnancy Outcome
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: underwent normal cesarean section without Postpartum hemorrhage after delivery
  Interventions: Procedure: Bilateral uterine artery ligation
- case group: cases underwent bilateral uterine artery ligation after Postpartum hemorrhage or Intrapartum hemorrhage after cesarean section.
  Interventions: Procedure: Bilateral uterine artery ligation

INTERVENTIONS:
Procedure: Bilateral uterine artery ligation — Bilateral UAL was done 2 cm under the Kerr incision (lower segment transverse). A 2-Vicryl absorbable suture (Ethicon, Neuilly-surSeine, France) was introduced from the anterior to posterior views of the myometrium 2-3 cm medial to the descending part of the uterine vessels within an avascular area in the broad ligament and tied. Following the surgery, the uterine tone and hemorrhage were managed.

SUMMARY:
The aim of this study is to assess the possible negative effects of uterine artery ligation on ovarian reserve markers and subsequent pregnancy outcomes

DETAILED DESCRIPTION:
One of the most common surgical methods for preserving fertility is uterine artery ligation. It is simple to do and effective at reducing Postpartum hemorrhage after delivery . Additionally, it is rather safe and permits future childbearing for the patients.

ELIGIBILITY:
Inclusion Criteria:

* 120 females aged from 20 to 35 years old
* with Postpartum hemorrhage or intrapartum hemorrhage after cesarean section
* did not respond to medical therapy
* performed successful bilateral uterine artery ligation for hemorrhage management.

Exclusion Criteria:

* The presence of male factor or tubal factor.
* Hypertension, autoimmune disease, morbid obesity, absence of lactation diabetes millets, vascular disease, smoking or the use of alcohol.
* The presence of additional surgery or medical disease.
* Detection of a uterine anomaly, history of intrauterine growth restriction in previous pregnancies.
* Usage of a hormonal therapy through the research.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females aged from 20 to 35 years old with Postpartum hemorrhage or intrapartum hemorrhage after cesarean section who did not respond to medical therapy and performed successful bilateral uterine artery ligation for hemorrhage management.
Study Population: Patients will be classified into two equal groups control group: underwent normal cesarean section without Postpartum hemorrhage, case group: cases underwent bilateral uterine artery ligation after Postpartum hemorrhage or intrapartum hemorrhage after cesarean section.
  All patients will be subjected to the following clinical parameters assessment (age, cycle history, body mass index, parity, preceding treatment and/or surgery menstruation characteristics (quantity of menstruation and dysmenorrhoea) and endometrial biopsy.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve by anti-mullerian hormone | 24 months after bilateral uterine artery ligation.
  Anti-mullerian hormone (AMH) level will be determined using a two-sided immunoassay that will be enzymatically amplified (ELISA). AMH was recorded at 6, 12 and 24 months after bilateral uterine artery ligation.

SECONDARY OUTCOMES:
Ovarian reserve by follicle stimulating hormone | 24 months after bilateral uterine artery ligation.
  follicle stimulating hormone (FSH) level will be determined using a two-sided immunoassay that will be enzymatically amplified (ELISA). FSH was recorded at 6, 12 and 24 months after bilateral uterine artery ligation.
Ovarian reserve by antral follicle counts | 24 months after bilateral uterine artery ligation.
  antral follicle counts were recorded at 6, 12 and 24 months after bilateral uterine artery ligation.
Percent of subsequent pregnancy cases | 24 months after bilateral uterine artery ligation.
  patients were asked about their desire for pregnancy in the future The data of subsequent pregnancy cases following bilateral UAL primary were recorded and follow-up was done at 6, 12 and 24 months after BUAL.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed M.E. Ossman, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the data will be available when requested
Supporting Information: Study Protocol, SAP
Time Frame: Available